CLINICAL TRIAL: NCT01585987
Title: A Randomized, Open-label, Two-arm Phase II Trial Comparing the Efficacy of Sequential Ipilimumab Versus Best Supportive Care Following First-line Chemotherapy in Subjects With Unresectable Locally Advanced/Metastatic Gastric or Gastro-esophageal Junction Cancer
Brief Title: An Efficacy Study in Gastric and Gastroesophageal Junction Cancer Comparing Ipilimumab Versus Standard of Care Immediately Following First Line Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA184-162; 2011-000853-22 (EudraCT Number)
Record Dates: First submitted 2012-04-25; First posted 2012-04-26 (Estimated); Results first posted 2015-11-18 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-04

CONDITIONS: Locally Advanced (Unresectable) or Metastatic Adenocarcinoma of the Gastric and Gastro-esophageal Junction
MeSH Terms: interventions — Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A: Ipilimumab (Experimental): Ipilimumab 10 mg/kg solution intravenously, 90 minute infusion, once every 3 weeks for 4 doses, then every 12 weeks until disease progression (for a maximum treatment period of 3 years from the first dose)
  Interventions: Biological: Ipilimumab
- Arm B: Best Supportive care (BSC) (Other): BSC may include the continuation of the Fluoropyrimidine that was used during the lead-in chemotherapy, but no other systemic anti cancer therapy
  Interventions: Other: Best Supportive care (BSC)

INTERVENTIONS:
Biological: Ipilimumab
  Other Names: BMS-734016
  Arms: Arm A: Ipilimumab
Other: Best Supportive care (BSC)
  Arms: Arm B: Best Supportive care (BSC)

SUMMARY:
The purpose of the study is to compare the efficacy of Ipilimumab and standard of care as sequential or maintenance treatment immediately after first-line chemotherapy in the treatment of unresectable or metastatic gastric and gastro-esophageal cancer.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com.

Key Inclusion Criteria:

* Histologically confirmed, unresectable locally advanced or metastatic adenocarcinoma of the gastric and gastro-esophageal junction
* Received first-line chemotherapy using fluoropyrimidine and platinum combination without disease progression
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Measurable disease by modified WHO criteria (unless complete response from previous chemotherapy)

Key Exclusion Criteria:

* Known Human Epidermal growth factor Receptor2 (HER2) positive status
* Radiological evidence of brain metastases
* History of severe autoimmune or immune mediated disease requiring prolonged immunosuppressive treatment
* Inadequate hematologic, renal and hepatic function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2012-07; Primary Completion 2014-07 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (30):
- United States (4):
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Nyu Clinical Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - The University Of Texas Md Anderson Cancer Center, Houston, Texas
- France (4):
  - Local Institution, Montpellier
  - Local Institution, Nice
  - Local Institution, Rennes
  - Local Institution, Toulouse
- Local Institution, Mainz, Germany
- Local Institution, Hong Kong, Hong Kong
- Italy (5):
  - Local Institution, Florence
  - Local Institution, Milan
  - Local Institution, Padua
  - Local Institution, Pisa
  - Local Institution, Roma
- Japan (4):
  - Local Institution, Nagoya, Aichi-ken
  - Local Institution, Saku-shi, Nagano
  - Local Institution, Osaka-sayama-shi, Osaka
  - Local Institution, Kitaadachi-gun, Saitama
- Poland (4):
  - Local Institution, Katowice, Ochojec
  - Local Institution, Krakow
  - Local Institution, Lodz
  - Local Institution, Olsztyn
- Local Institution, Moscow, Russia
- Local Institution, Singapore, Singapore
- South Korea (2):
  - Local Institution, Gyeonggi-do
  - Local Institution, Seoul
- Spain (2):
  - Local Institution, Barcelona
  - Local Institution, Madrid
- Local Institution, Taipei, Taiwan

REFERENCES:
- [Derived] Chang X, Ge X, Zhang Y, Xue X. The current management and biomarkers of immunotherapy in advanced gastric cancer. Medicine (Baltimore). 2022 May 27;101(21):e29304. doi: 10.1097/MD.0000000000029304. PMID 35623069
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Acceptable first-line chemotherapy before randomization to this study for a participant was a regimen containing a fluoropyrimidine agent and a platinum salt. Study initiated July 2012. Primary endpoint July 2014. Study completed April 2015.
Pre-assignment Details: 114 enrolled and randomized. 29 enrolled but not randomized to treatment group: 26 no longer met study criteria; 2 withdrew consent, 1 other.
Groups:
- Ipilimumab: Ipilimumab 10 milligram per kilogram body weight (mg/kg) solution intravenously (IV), over 90 minutes, once every 3 weeks for 4 doses, then 10 mg/kg every 12 weeks until disease progression (for a maximum treatment period of 3 years from the first dose). The option of re-introduction, defined as an additional 4 doses of ipilimumab (a dose of 10 mg/kg every 3 weeks) was allowed only at discretion of the investigator if criteria for re-induction were met.
- All Best Supportive Care (BSC): All BSC includes both active and non-active BSC. Active BSC includes the continuation of the fluoropyrimidine that was used during the lead-in chemotherapy (prior to randomization to this study), but no other active systemic anti-cancer treatment. In non-active BSC, the fluoropyrimidine used during lead-in chemotherapy was not continued on study and no other chemotherapy or active treatment was used
Period: Randomized
Arm/Group | Ipilimumab | All Best Supportive Care (BSC)
Started | 57 | 57
Completed | 57 | 51
Not Completed | 0 | 6
Not completed — Withdrawal by Subject | 0 | 4
Not completed — No longer met criteria | 0 | 2
Period: Treated
Arm/Group | Ipilimumab | All Best Supportive Care (BSC)
Started | 57 | 51
Completed | 3 | 2
Not Completed | 54 | 49
Not completed — Disease Progression | 39 | 36
Not completed — Study Drug Toxicity | 9 | 5
Not completed — Adverse Event | 3 | 0
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Maximum Clinical Benefit | 0 | 1
Not completed — Non-Specified | 1 | 2
Not completed — Subject Request | 0 | 1
Not completed — Poor/Non-Compliance | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants randomized to a treatment arm are summarized.
Groups:
- All Best Supportive Care (BSC): BSC may include the continuation of the fluoropyrimidine that was used during the lead-in chemotherapy (prior to randomization to this study), but no other active systemic anti-cancer treatment.
- Total: Total of all reporting groups
Arm/Group | Ipilimumab | All Best Supportive Care (BSC) | Total
Number analyzed (Participants) | 57 | 57 | 114
Age, Continuous [Median (Full Range); unit: years] | 65.0 [34 to 86] | 62.0 [32 to 80] | 64.0 [32 to 86]
Age, Customized [Number; unit: participants]
  Less than (<) 65 years of age | 28 | 35 | 63
  Greater, equal to (>=) 65 years of age | 29 | 22 | 51
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 16 | 37
  Male | 36 | 41 | 77
Region of Enrollment [Number; unit: participants]
  Russian Federation | 1 | 1 | 2
  Singapore | 1 | 1 | 2
  Hong Kong | 1 | 0 | 1
  United States | 8 | 6 | 14
  Japan | 7 | 5 | 12
  Taiwan | 1 | 0 | 1
  Poland | 0 | 2 | 2
  Korea, Republic of | 21 | 24 | 45
  Italy | 11 | 8 | 19
  France | 3 | 5 | 8
  Germany | 1 | 0 | 1
  Spain | 2 | 5 | 7

OUTCOME MEASURES:

1. Primary Outcome: Immune-related Progression Free Survival (irPFS) as Per Assessment of a Blinded Independent Review Committee (IRC) According to Immune Related Response Criteria (irRC) Guidelines
Description: irPFS is defined as the time between the randomization date and the time of disease progression per irRC or death, whichever occurs first. irRC criteria=Measurable new lesions: incorporated into the tumor burden (eg, added to the index lesions); do not define progression unless the total measurable tumor burden increases by the required amount (25%). New non-measurable lesions: not considered progression if the total measurable tumor burden is stable or shrinking. irPFS was measured in months.
Time Frame: Randomization up to 91 irPFS events (Approximately 19 months )
Population: All participants who were randomized were summarized.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- All Best Supportive Care (BSC): BSC may include the continuation of the fluoropyrimidine that was used during the lead-in chemotherapy (prior to randomization to this study), but no other active systemic anti-cancer treatment. All BSC = Active and non-active BSC.
Arm/Group | Ipilimumab | All Best Supportive Care (BSC)
Number analyzed (Participants) | 57 | 57
Months | 2.9240 [1.6100 to 5.1580] | 4.8950 [3.4500 to 6.5380]
Statistical Analysis 1: Comparison: Ipilimumab vs All Best Supportive Care (BSC); Test type: Superiority or Other; p = 0.0972, Log Rank — Significance level used: 0.2; Hazard Ratio (HR) = 1.439, 80% CI 2-sided [1.085 to 1.908] — The hazard ratio and its associated two-sided 80% confidence interval (CI) was estimated via a stratified Cox model with treatment arm as the only covariate in the model

2. Secondary Outcome: Progression Free Survival (PFS) Per Modified World Health Organization (mWHO) Criteria
Description: PFS per mWHO was defined as the time between the randomization date and the time of disease progression per mWHO criteria or death, whichever occurred first and was measured in months. mWHO criteria: New lesions always mean progression; Changes in non-measurable lesions contribute in the definitions of Complete Response (CR), Partial Response (PR), Stable Disease (SD) and Progressive Disease (PD).
Time Frame: Randomization up to 91 irPFS events (Approximately 19 months )
Population: All participants randomized to a treatment group were summarized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ipilimumab | All Best Supportive Care (BSC)
Number analyzed (Participants) | 57 | 57
Months | 2.7270 [1.4460 to 2.9570] | 4.8950 [3.4500 to 6.0780]
Statistical Analysis 1: Comparison: Ipilimumab vs All Best Supportive Care (BSC); Test type: Superiority or Other; p = 0.0336, Log Rank — Significance level used: 0.2; Hazard Ratio (HR) = 1.588, 80% CI 2-sided [1.199 to 2.103]

3. Secondary Outcome: Overall Survival (OS) at Primary Endpoint
Description: OS was defined as the time from the date of randomization until the date of death. For those participants who have not died, OS was censored on the last date the participant was known to be alive.
Time Frame: Randomization up to 91 irPFS events (Approximately 19 months)
Population: All participants randomized to a treatment group and who received at least one dose of active drug were summarized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ipilimumab | All Best Supportive Care (BSC)
Number analyzed (Participants) | 57 | 51
Months | 16.7560 [11.7950 to 23.1290] | 12.0570 [9.3310 to NA] — Not estimable since the largest observation was censored.
Statistical Analysis 1: Comparison: Ipilimumab vs All Best Supportive Care (BSC); Test type: Superiority or Other; p = 0.6433, Log Rank — Significance level used: 0.2; Hazard Ratio (HR) = 0.874, 80% CI 2-sided [0.602 to 1.269] — HR was based on a stratified Cox proportional hazards model with treatment arm as the only covariate in the model

4. Secondary Outcome: Overall Survival (OS) at Study Completion
Description: as for outcome 3
Time Frame: Randomization up to end of study, April 2015 (Approximately 28 months)
Population: All participants randomized to a treatment group and who received at least one dose of active drug were summarized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ipilimumab | All Best Supportive Care (BSC)
Number analyzed (Participants) | 57 | 57
Months | 12.68 [10.51 to 18.92] | 12.06 [9.33 to NA] — Upper limit was not estimable.

5. Secondary Outcome: Percentage of Participants With Immune-Related Best Overall Response (irBOR)
Description: IrBOR rate was defined as the number of participants whose Immune-related Best Overall Response (irBOR) criteria was Immune-related Complete Response (irCR) or Immune-related Partial Response (irPR), divided by the total number of participants. The immune-related sum of products of diameters (irSPD) incorporates - in addition to the index lesions - measurable new lesions that may have developed on-study, providing an assessment that includes both index and new lesions. irCR=Complete disappearance of all tumor lesions (both index and non-index lesions with no new measurable/unmeasurable lesions). irPR=A 50% or greater decrease, relative to baseline of the irSPD, (based on irSPD of all index lesions and any measurable new lesions).
Time Frame: Randomization up to 91 irPFS events (Approximately 19 months)
Population: All participants randomized to a treatment group were summarized.
Measure: Number; unit: percentage of participants
Arm/Group | Ipilimumab | All Best Supportive Care (BSC)
Number analyzed (Participants) | 57 | 57
percentage of participants | 1.8 | 7.0
Statistical Analysis 1: Comparison: Ipilimumab vs All Best Supportive Care (BSC); Test type: Superiority or Other; p = 0.3686, Cochran-Mantel-Haenszel — Significance level used: 0.2; Odds Ratio (OR) = 4.0549, 80% CI 2-sided [0.7009 to 47.6447]

ADVERSE EVENTS:
Time Frame: Randomization to end of study (April 2015)
Description: Study initiated: July 2012; End of Study: April 2015
Groups:
- Active Best Supportive Care (BSC): Active BSC includes the continuation of the fluoropyrimidine that was used during the lead-in chemotherapy (prior to randomization)
- Non-Active BSC: Non-Active BSC involves supportive care with cessation of chemotherapy (no active drug)
Arm/Group | Ipilimumab | Active Best Supportive Care (BSC) | Non-Active BSC
Serious Adverse Events (participants affected / at risk) | 31/57 | 19/45 | 1/6
Other Adverse Events (participants affected / at risk) | 55/57 | 42/45 | 4/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ipilimumab (N=57) | Active Best Supportive Care (BSC) (N=45) | Non-Active BSC (N=6)
Abdominal pain (Gastrointestinal disorders) | 1 | 4 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 7 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 1
Transaminases increased (Investigations) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypopituitarism (Endocrine disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Obstruction gastric (Gastrointestinal disorders) | 0 | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 0
Cholecystocholangitis (Hepatobiliary disorders) | 1 | 0 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 2 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypothermia (General disorders) | 1 | 0 | 0
Performance status decreased (General disorders) | 1 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Death (General disorders) | 1 | 0 | 0
Device related infection (Infections and infestations) | 1 | 0 | 0
Disease progression (General disorders) | 6 | 4 | 0
Endocrine disorder (Endocrine disorders) | 1 | 0 | 0
General physical health deterioration (General disorders) | 1 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 0
Colitis (Gastrointestinal disorders) | 3 | 0 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 0
Escherichia sepsis (Infections and infestations) | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Malaise (General disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Pneumonia (Infections and infestations) | 4 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 3 | 2 | 0
Asthenia (General disorders) | 1 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0
Compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Hepatitis acute (Hepatobiliary disorders) | 1 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Abdominal infection (Infections and infestations) | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 7 | 0 | 0
Fatigue (General disorders) | 3 | 1 | 0
Gastrointestinal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ipilimumab (N=57) | Active Best Supportive Care (BSC) (N=45) | Non-Active BSC (N=6)
Abdominal pain (Gastrointestinal disorders) | 12 | 16 | 0
Alanine aminotransferase increased (Investigations) | 9 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 21 | 14 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0
Pyrexia (General disorders) | 9 | 7 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 5 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 1 | 0
Pain (General disorders) | 3 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 4 | 8 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 25 | 3 | 0
Abdominal pain upper (Gastrointestinal disorders) | 6 | 4 | 0
Aspartate aminotransferase increased (Investigations) | 9 | 2 | 0
Constipation (Gastrointestinal disorders) | 10 | 12 | 0
Dizziness (Nervous system disorders) | 5 | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 8 | 2 | 0
Hypothyroidism (Endocrine disorders) | 4 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 6 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 15 | 2 | 1
Weight decreased (Investigations) | 11 | 5 | 0
Dyspepsia (Gastrointestinal disorders) | 5 | 3 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 1 | 0
Nausea (Gastrointestinal disorders) | 19 | 16 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 7 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 4 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 3 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 2 | 0
Influenza like illness (General disorders) | 0 | 3 | 0
Vomiting (Gastrointestinal disorders) | 17 | 12 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 2 | 0
Haemoglobin decreased (Investigations) | 3 | 1 | 0
Weight increased (Investigations) | 3 | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 12 | 5 | 0
Anxiety (Psychiatric disorders) | 0 | 4 | 0
Asthenia (General disorders) | 12 | 7 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Chest pain (General disorders) | 3 | 1 | 0
Chills (General disorders) | 3 | 1 | 0
Headache (Nervous system disorders) | 4 | 1 | 0
Insomnia (Psychiatric disorders) | 5 | 6 | 0
Oedema peripheral (General disorders) | 8 | 5 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1
Abdominal distension (Gastrointestinal disorders) | 3 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 6 | 0
Diarrhoea (Gastrointestinal disorders) | 19 | 9 | 0
Fatigue (General disorders) | 26 | 9 | 0
Hypertension (Vascular disorders) | 2 | 2 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 5 | 5 | 0
Mucosal inflammation (General disorders) | 0 | 4 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 10 | 7 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.